CLINICAL TRIAL: NCT02353728
Title: Detection, Monitoring, and Molecular Characterization of Leukemic Stem Cells From Patients With Chronic Myeloid Leukemia (CML) Undergoing Therapy With Nilotinib
Brief Title: Stem Cell Monitoring for CML Patients Undergoing Nilotinib Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1403014950
Record Dates: First submitted 2015-01-13; First posted 2015-02-03 (Estimated); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Patients (Experimental): Nilotinib at a dose of 300 mg P.O. twice a day (BID) daily
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib
  Other Names: Tasigna; AMN107

SUMMARY:
The study is an open-label phase 2 clinical and translational trial designed to evaluate the effects of nilotinib on the leukemic stem cell population in subjects with newly diagnosed chronic phase chronic myeloid leukemia (Ph+ CML in CP). Nilotinib is FDA-approved to treat subjects with Ph+ CML in CP. Subjects on study will be monitored according to accepted National Cancer Comprehensive Network [NCCN] clinical guidelines for 24 months. After 24 months, if continued therapy is needed subjects will be transitioned to commercial supply of study drug.

DETAILED DESCRIPTION:
Patients with newly diagnosed Ph+ CML in chronic phase will be eligible for enrollment in this trial. Prior treatment with nilotinib for less than 2 weeks and hydroxyurea is allowed.

Before therapy and during therapy, peripheral blood and bone marrow samples will be obtained for cytogenetic and molecular evaluations. During study, blood will be collected at approximately month 1, month 3, and every 3 months thereafter; aspirate samples will be collected at approximately month 1, month 3, and month 12. These samples will be collected to analyze the quantitative and qualitative changes in the leukemic stem cell population before and during therapy with nilotinib. The study is intended as a hypothesis finding analysis in order to establish whether in response to nilotinib therapy, defined differences in the baseline or therapy-induced changes in the characteristics of the stem cell population will be predictive of the ability to successfully discontinue therapy in subjects with CML.

In order to determine the effect of nilotinib in stem and progenitor populations we will evaluate 40 newly diagnosed CML subjects undergoing treatment with nilotinib at different time points. We will evaluate the levels of expression of Breakpoint Cluster Region-Abelson protooncogene (BCR-ABL) in purified stem cell populations during the course of treatment. In addition, we will compare the stem and progenitor populations present during the course of treatment in peripheral blood and bone marrow. We will perform transcriptional profiling of such populations to determine changes in signaling pathways driving survival, self-renewal or proliferation. Whole exome sequencing will be also performed in all diagnostic samples to determine whether there are novel cooperating mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. Eastern Cooperative Oncology Group (ECOG) Performance status 0,1, or 2
3. Documented diagnosis of Ph+ Chronic phase CML:

   * Chronic phase: None of the criteria for accelerated or blastic phase
   * Accelerated phase

     1. Blasts ≥ 15% in blood or BM
     2. Blasts plus progranulocytes ≥ 30% in blood or bone marrow (BM)
     3. Basophilia ≥ 20% in blood or BM
     4. Platelets < 100 × 109/L unrelated to therapy
     5. Cytogenetic clonal evolution
   * Blast phase

     1. ≥ 30% blasts in blood or BM
     2. Extramedullary disease with localized immature blasts
4. Adequate end organ function, defined as the following:

   * Creatinine < 1.5 x upper limit of normal (ULN)
   * Absolute neutrophil count (ANC) > 1.5 x 109/L
   * Platelets > 100 x 109/L
   * Total bilirubin < 1.5 x ULN (Does not apply to patients with isolated hyperbilirubinemia [e.g., Gilbert's disease] grade <3)
   * Aspartate aminotransferase (AST) (SGOT) and Alanine aminostransferase (ALT) (SGPT) < 3 x ULN
   * Serum amylase and lipase ≤ 2 x ULN
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Patients must have the following laboratory values (WNL = within normal limits at the local institution lab) or corrected to within normal limits with supplements prior to the first dose of study medication:

     1. Potassium (WNL)
     2. Magnesium (WNL)
     3. Phosphorus (WNL)
     4. Calcium (WNL)

Exclusion Criteria:

1. Previous treatment with any other tyrosine kinase inhibitor except for up to 2 weeks of nilotinib
2. Impaired cardiac function including any one of the following:

   * Inability to monitor the QT interval on ECG
   * Congenital long QT syndrome or a known family history of long QT syndrome.
   * Clinically significant resting brachycardia (<50 beats per minute)
   * Q-T Corrected (corrected Q-T interval) (QTc) > 450 msec on baseline ECG. If QTc >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
   * Myocardial infarction within 12 months prior to starting study Other clinically significant uncontrolled heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension)
   * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
   * Complete left bundle branch block
   * Right bundle branch block plus left anterior/posterior hemiblock
   * Use of ventricular-paced pacemaker
   * History of unstable angina within 1 year of study entry
3. Patients currently receiving treatment with strong CYP3A4 inhibitors and treatment cannot be either discontinued or switched to a different medication prior to starting study drug. (http://medicine.iupui.edu/clinpharm/ddis/) ).
4. Patients currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug (http://crediblemeds.org/)
5. Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection or gastric bypass surgery).
6. History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
7. Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes, uncontrolled infection)
8. History of another active malignancy within 5 years prior to study entry with the exception of previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively
9. Known presence of significant congenital or acquired bleeding disorder unrelated to cancer
10. Major surgery within 4 weeks prior to Day 1 of the study or who have not recovered from prior surgery
11. Treatment with other investigational agents within 30 days of Day 1.
12. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of female after conception and until the termination of gestation, confirmed by a positive Human chorionic gonadotropin (hCG) laboratory test. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during the study and for 14 days after the final dose of nilotinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen K Ritchie, MD, Principal Investigator — Associate Professor of Clinical Medicine
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Nilotinib at a dose of 300 mg P.O. twice a day (BID) daily
  Nilotinib
Period: Overall Study
Arm/Group | All Patients
Started | 16
Completed | 15
Not Completed | 1
Not completed — Subject non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Leukemic Stem Cells Present in Bone Marrow Aspirate Samples, in This Patient Population
Description: The data obtained from these bone marrow samples, from these patients, may identify stem cell variables that can more accurately predict the success of discontinuation of tyrosine kinase inhibitor (TKI) therapy.
Time Frame: 1 month, 3 months, 12 months
Population: 16 patients were treated, 7 patients were not evaluable due to bone marrow samples not being available. Not all timepoints for each patient are reported due to bone marrow samples not being available. Bone marrow samples were not available due to: samples not being collected from a bone marrow procedure; bone marrow procedures not being performed so no sample could be obtained; or collected or sample was not evaluable.
Measure: Number; unit: percentage of leukemic stem cells
Arm/Group | All Patients
Number analyzed (Participants) | 9
percentage of leukemic stem cells
  WCMC-007 (3 months): number analyzed (Participants) | 1
  WCMC-007 (3 months) | 37.4
  WCMC-010 (1 month): number analyzed (Participants) | 1
  WCMC-010 (1 month) | 2.32
  WCMC-011 (12 months): number analyzed (Participants) | 1
  WCMC-011 (12 months) | 0.7
  WCMC-013 (1 month): number analyzed (Participants) | 1
  WCMC-013 (1 month) | 7.04
  WCMC-013 (12 months): number analyzed (Participants) | 1
  WCMC-013 (12 months) | 24.2
  WCMC-014 (1 month): number analyzed (Participants) | 1
  WCMC-014 (1 month) | 9.57
  WCMC-014 (3 month): number analyzed (Participants) | 1
  WCMC-014 (3 month) | 14.6
  WCMC-014 (12 months): number analyzed (Participants) | 1
  WCMC-014 (12 months) | 5.37
  WCMC-015 (1 month): number analyzed (Participants) | 1
  WCMC-015 (1 month) | 10.9
  WCMC-015 (3 months): number analyzed (Participants) | 1
  WCMC-015 (3 months) | 4.33
  WCMC-017 (1 month): number analyzed (Participants) | 1
  WCMC-017 (1 month) | 10.9
  WCMC-017 (3 month): number analyzed (Participants) | 1
  WCMC-017 (3 month) | 13.7
  WCMC-020 (3 months): number analyzed (Participants) | 1
  WCMC-020 (3 months) | 11.7
  WCMC-020 (12 months): number analyzed (Participants) | 1
  WCMC-020 (12 months) | 19.3
  WCMC-021 (3 month): number analyzed (Participants) | 1
  WCMC-021 (3 month) | 3.67

ADVERSE EVENTS:
Time Frame: Up to 5 years and 6 months.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 5/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=16)
Abdominal pain/vomiting/nausea (Gastrointestinal disorders) | 1 (1)
Diarrheal illness (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Intermittent left upper quadrant pain (General disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Livido reticularis (Skin and subcutaneous tissue disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=16)
Abdominal discomfort (pain or cramps) (Gastrointestinal disorders) | 5 (10)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
ALT elevated (Investigations) | 4 (4)
ALP elevated (Investigations) | 5 (7)
Allergic rhinitis (Immune system disorders) | 1 (1)
Amylase increased (Investigations) | 2 (3)
Anemia (Investigations) | 11 (18)
Chest pain/tightness (General disorders) | 5 (8)
Anxiety (Psychiatric disorders) | 2 (2)
Appetite change (Gastrointestinal disorders) | 2 (2)
AST increased (Investigations) | 3 (3)
Back pain (General disorders) | 1 (1)
Basophilia (Investigations) | 1 (1)
Headaches (Nervous system disorders) | 5 (6)
Pain - knee (General disorders) | 3 (3)
Bilirubin elevated (Investigations) | 2 (9)
Rash (Skin and subcutaneous tissue disorders) | 7 (16)
Breasts cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Bradycardia (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Cold/cold symptoms (General disorders) | 4 (5)
Chipped tooth (General disorders) | 1 (1)
Elevated cholesterol (Investigations) | 4 (4)
Hyperglycemia (Investigations) | 5 (19)
Hyperlipidemia (Investigations) | 3 (3)
Nasal discharge (General disorders) | 1 (1)
Conjunctiva injected (Eye disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
COVID/COVID Symptoms (Infections and infestations) | 2 (2)
Diabetes (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Dizziness/Lightheadedness (General disorders) | 2 (2)
Dog bite (General disorders) | 1 (1)
Dry/Red eyes (Eye disorders) | 5 (6)
Dry mouth/perioral dryness (General disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Elevated TSH (Investigations) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 2 (2)
Fall (General disorders) | 1 (1)
Fatigue (General disorders) | 10 (14)
Fever (General disorders) | 3 (4)
Folliculitis (Skin and subcutaneous tissue disorders) | 2 (4)
Gastric reflux syndrome (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Generalized pain (General disorders) | 3 (3)
Hair darkening (General disorders) | 1 (1)
Hair thinning (General disorders) | 1 (2)
Heart burn (Gastrointestinal disorders) | 2 (2)
Hematocrit decreased (Investigations) | 1 (1)
Hemoglobin decrease (Investigations) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypocalcemia (Investigations) | 4 (12)
Hypoalbunemia (Investigations) | 1 (1)
Hypoglycemia (Investigations) | 2 (2)
Hyponatremia (Investigations) | 2 (2)
Hypophosphatemia (Investigations) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Intermittent foul breath (Gastrointestinal disorders) | 1 (1)
Iron deficiency (Investigations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Hand/wrist pain (General disorders) | 2 (2)
Rib pain (General disorders) | 2 (2)
Lesion (General disorders) | 2 (2)
Leukocytosis (Investigations) | 5 (5)
Leukopenia (Investigations) | 6 (11)
Low MCV (Investigations) | 1 (1)
Lipase increased (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 3 (9)
Mid renal insufficiency (Renal and urinary disorders) | 1 (1)
Missed period (Reproductive system and breast disorders) | 1 (1)
Moles (Skin and subcutaneous tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neutropenia (Investigations) | 5 (8)
Night sweats (General disorders) | 1 (1)
Overweight (Metabolism and nutrition disorders) | 1 (1)
Leg/Knee pain (General disorders) | 3 (3)
Pain at needle entry site (Injury, poisoning and procedural complications) | 2 (2)
Pain with urination (Renal and urinary disorders) | 1 (1)
Palpable spleen (General disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (6)
Periorbital edema (Eye disorders) | 1 (1)
Thrombocytopenia (Investigations) | 10 (25)
Platelet count increased (Investigations) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Restless legs (Nervous system disorders) | 1 (1)
Broken/fractured arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Heel pain (General disorders) | 1 (1)
Neck pain (General disorders) | 1 (1)
Ringing in ears (Ear and labyrinth disorders) | 1 (1)
Scalp irritation/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Seasonal allergies (Immune system disorders) | 1 (1)
Scalp nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seborrheic Keratoses (Skin and subcutaneous tissue disorders) | 1 (1)
Sensation of bugs crawling on left shoulder (General disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Splenic pain (General disorders) | 1 (2)
Stomach pain (General disorders) | 2 (2)
Stomach virus (Infections and infestations) | 1 (1)
Strep throat (Infections and infestations) | 1 (1)
Swelling of upper lip (General disorders) | 1 (1)
Tenderness behind knees (Musculoskeletal and connective tissue disorders) | 1 (1)
Toothache (General disorders) | 1 (1)
Upper respiratory infection/symptoms (Infections and infestations) | 3 (4)
Uric acid elevated (Investigations) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight gain (Metabolism and nutrition disorders) | 2 (2)
Yeast infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02353728/Prot_SAP_000.pdf